CLINICAL TRIAL: NCT01502436
Title: An Exploration of the Relationship Between Chronic Pain and Suicide Attempt Among Veterans
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 06-0214
Record Dates: First submitted 2011-12-28; First posted 2011-12-30 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Posttraumatic Stress Disorder; Traumatic Brain Injury; Suicide Attempt
Keywords: posttraumatic stress disorder; traumatic brain injury; Suicide Attempt; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the relationship between attempted and/or completed suicide and reported experience of chronic pain among an adult veteran population. Specific aims include a) examining the experience of chronic pain between patients who have either attempted and/or completed suicide, non-suicide attempt mental health patients, and non-mental health chronic pain patients and b) determining possible differences in reported experiences of chronic pain based on mental and physical diagnoses, age, gender, ethnicity, occupation, and patient's recorded perceptions of depression and/or quality of life. As articulated in the Amendment approved on June 13, 2008, additional areas of interest include histories of neurological disease (e.g. traumatic brain injury) and/or mental health diagnoses. History of both neurologic disease and mental health diagnoses will also be identified by chart review (per approval obtained June 13, 2008). As such this study will also compare differences (e.g., mental health, neurological disease) between veterans who have history of a suicide attempt, completion, or a lifetime history of suicidality and matched control veterans without a history of suicide attempts, completions, or lifetime history of suicide. The relationship between suicidal behavior, attempted/completed suicide, and reported Post Traumatic Stress Disorder (PTSD) symptoms among an adult veteran population is also of interest. Additionally, this data set will be used to complete a validation study regarding the Self-Directed Violence Classification System (SDVCS). Specifically, relevant information in subject chart notes regarding self-directed violence (SDV) will be used to categorize thoughts and behaviors according to the SDVCS.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Record of a suicide attempt or completion between October 2004 and February 2006

Exclusion Criteria:

* For cases: upon chart review, no record of a suicide attempt or completion within the specified time frame

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans who received care in the VA.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, PhD, Principal Investigator — VA VISN 19 MIRECC
Locations (1):
- Eastern Colorado Healthcare System, Denver, Colorado, United States